CLINICAL TRIAL: NCT05028140
Title: National, Multicenter, Randomized, Double-blind, Triple-dummy, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Piemonte Association in the Treatment of Type II Diabetes Mellitus
Brief Title: Efficacy and Safety of Piemonte Association in the Treatment of Type II Diabetes Mellitus
Acronym: PIEMONTE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS1020 - PIEMONTE
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Type II Diabetes
Keywords: Type II diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Piemonte association (Experimental): The study is triple-dummy, thus the patient must take 3 tablets once a day, as follows:
  1 tablet Piemonte, oral;
  1 placebo tablet of empagliflozin, oral;
  1 placebo tablet of piglitazone, oral.
  Interventions: Drug: PIEMONTE; Other: PLACEBO EMPAGLIFLOZIN; Other: PLACEBO PIOGLITAZONE
- Empagliflozin (Active Comparator): The study is triple-dummy, thus the patient must take 3 tablets once a day, as follows:
  1 placebo tablet of Piemonte, oral;
  1 tablet of empagliflozin, oral;
  1 placebo tablet of piglitazone, oral.
  Interventions: Other: PIEMONTE PLACEBO; Drug: EMPAGLIFLOZIN; Other: PLACEBO PIOGLITAZONE
- Pioglitazone (Active Comparator): The study is triple-dummy, thus the patient must take 3 tablets once a day, as follows:
  1 placebo tablet of Piemonte, oral;
  1 placebo tablet of empagliflozin, oral;
  1 tablet of piglitazone, oral.
  Interventions: Other: PIEMONTE PLACEBO; Other: PLACEBO EMPAGLIFLOZIN; Drug: PIOGLITAZONE

INTERVENTIONS:
Drug: PIEMONTE — Piemonte association 1 coated tablet once a day
  Arms: Piemonte association
Other: PIEMONTE PLACEBO — Placebo of Piemonte association 1 coated tablet once a day
  Arms: Empagliflozin; Pioglitazone
Drug: EMPAGLIFLOZIN — Empagliflozin 25 mg 1 coated tablet once a day
  Arms: Empagliflozin
Other: PLACEBO EMPAGLIFLOZIN — Placebo of empagliflozin 25 mg 1 coated tablet once a day
  Arms: Piemonte association; Pioglitazone
Drug: PIOGLITAZONE — Pioglitazone 30 mg 1 tablet once a day
  Arms: Pioglitazone
Other: PLACEBO PIOGLITAZONE — Placebo of pioglitazone 30 mg 1 tablet once a day
  Arms: Empagliflozin; Piemonte association

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Piemonte association in the treatment of type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the consent form;
* Diagnosis of type II diabetes mellitus, and who did not reach the therapeutic goal of HbA1c with previous dietary, physical exercise, and previous therapies at stable doses within 3 months.

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of participants;
* History of alcohol abuse or illicit drug use;
* Participation in a clinical trial in the year prior to this study;
* Pregnancy or risk of pregnacy and lactating participants;
* Known hypersensitivity to any of the formula compounds;
* Type 1 diabetes.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin | 120 days
  Change from baseline in glycated hemoglobin

SECONDARY OUTCOMES:
Adverse events | 150 days
  Incidence and severity of adverse events recorded during the study

CONTACTS AND LOCATIONS:
Locations (1):
- EMS, Hortolândia, São Paulo, Brazil